CLINICAL TRIAL: NCT02628938
Title: Effect of Miswak and Miswak Extract on Oral Malodor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Riyadh Colleges of Dentistry and Pharmacy (Other)
Responsible Party: Principal Investigator, Mohammad Ramadan Rayyan, Assistant professor, Riyadh Colleges of Dentistry and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUGRP/2013/114
Record Dates: First submitted 2015-12-07; First posted 2015-12-11 (Estimated); Results first posted 2016-05-11 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-04

CONDITIONS: Oral Malodor; Halitosis
Keywords: Halitosis; Oral Malodor; Miswak; Salvadora Persica
MeSH Terms: conditions — Halitosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Miswak extract mouth wash (Experimental): 50% mouthwash aqueous solution 5ml twice a day for 7 days
  Interventions: Other: Miswak extract mouth wash
- Miswak sticks (Experimental): Sticks twice a day for 7 days
  Interventions: Other: Miswak stick
- Chlorohexidine gluconate mouth wash (Active Comparator): 0.2% mouth wash aqueous solution (Oraxine ®) 5 ml twice a day for 7 days
  Interventions: Other: Chlorohexidine gluconate

INTERVENTIONS:
Other: Miswak extract mouth wash — 50% Miswak extract mouth wash (5ml) twice a day for 7 days
  Other Names: Salvadora persica mouth wash
  Arms: Miswak extract mouth wash
Other: Miswak stick — Miswak stick twice a day for 7 days
  Arms: Miswak sticks
Other: Chlorohexidine gluconate — 5 ml of 0.2% Chlorohexidine gluconate mouth wash Oraxine ® twice a day for 7 days
  Other Names: Oraxine ®
  Arms: Chlorohexidine gluconate mouth wash

SUMMARY:
The aim of this experiment is to investigate the effect of Miswak on oral malodor and to determine whether this effect -if present- is the result of the mechanical action of Miswak or the chemical effect of its extract

DETAILED DESCRIPTION:
The study was designed as a randomized, parallel group clinical trial with one control and two test groups. The efficacy of each modality was evaluated by comparing the oral malodor indicators before use with those after 15 minutes (masking effect) and 7 days (therapeutic effect) of use. Three indicators for oral malodor were recorded; Organoleptic scores (OLS), Self-assessment of oral malodor, and the level of volatile sulfur compounds (VSC) measured by a breath checker device.

Ethical committee approval was obtained from the research center in Riyadh Colleges of Dentistry and Pharmacy (FUGRP/2013/114) prior to conducting of the study.

Between March and December 2014, screening of volunteered 212 female dental students aged 18-35 years was carried out. Preliminary interview and clinical examinations were done for all volunteers to select the sample according to the study inclusion and exclusion criteria. To be included in the study, the participants should report that they suffered from bad oral malodor and also should have an organoleptic score of 2 or above. Total of 167 interviewed subjects were excluded from the study for not fulfilling the eligibility criteria and a final sample size of 45 volunteers who have satisfied the criteria were selected in the study. The objectives of the study were fully explained and an informed written consent was obtained to participate in the study.

One week before the baseline readings all the 45 participants received instructions to avoid eating spicy foods, garlic and onions 2 days prior to the assessment. All participants were instructed to maintain their current oral hygiene regime.

The included participants (N=45) were randomly divided into 3 groups. (Group ME): 15 participants were asked to rinse with 50% Miswak extract mouth wash (5ml) twice a day for 7 days. Each participant was given a determined volume of the mouth wash and a marked scoop for the prescribed dose. Compliance of the participants was checked by measuring the remaining volume in the bottle during the second visit.

(Group MS): 15 participants were taught and instructed to use Miswak stick twice a day for 7 days. Length of the Miswak stick was measured on the second visit to assess the compliance of the participants in using them.

(Group CH): 15 participants were taught and instructed to rinse with 5 ml of 0.2% Chlorohexidine gluconate mouth wash (Oraxine ®) twice a day for 7 days. Each participant was given a determined volume of the mouth wash and a marked scoop for the prescribed dose. Compliance of the participants was checked by measuring the remaining volume in the bottle during the second visit.

To prepare the Miswak extract, a group of fresh Miswak sticks were collected from the local market and chopped into very small pieces. The sticks were then allowed to dry in room temperature for 2 days before they were ground into powder. To prepare the mouth wash, 10 gm of the powder was added to 100 ml of sterile distilled water and allowed to soak for another two days at a temperature of 4°C. It was then centrifuged for 15 minutes at 2000 rpm and then filtered using 0.45 μm pore size paper. The resultant solution was further diluted by distilled water by the ratio of 1:1 and used within one week.

Measurements of oral malodor indicators:

All readings were taken early in the morning one to three hours after breakfast and tooth brushing. Measurements included the following:

* Self-assessment of mouth odor
* Organoleptic scores (OLS)
* Volatile sulfur compound

Data analysis was performed using paired t-test to compare the different indicator scores before and after the use of each method. One way ANOVA was also performed to test the significance of the difference between the three methods in reducing oral malodor. A P<0.05 was accepted as the level of significance.

ELIGIBILITY:
Inclusion Criteria:

* the participants should report that they suffered from bad oral malodor
* organoleptic score of 2 or above

Exclusion Criteria:

* smoking
* current systemic diseases or medical treatment
* active caries or any faulty restorations
* acute sinusitis or oro-pharyngeal infection
* chronic periodontitis
* pregnancy
* breast feeding
* eating very spicy food
* use of antibiotic during the last two months before the start of the study

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 212 (Actual)
Dates: Start 2014-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad R Rayyan, MDS, Principal Investigator — Assistant professor
Locations (1):
- Riyadh colleges of dentistry and pharmacy, Riyadh, Riyadh Region, Saudi Arabia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place between March and December 2014 in the dental clinics of Riyadh colleges of Dentistry and Pharmacy
Pre-assignment Details: 212 female students aged 18-35 were screened. 167 were excluded for not meeting the inclusion criteria. Only 45 were finally enrolled and distributed on the three groups
Period: Overall Study
Arm/Group | Miswak Extract Mouth Wash | Miswak Sticks | Chlorohexidine Gluconate Mouth Wash
Started | 15 | 15 | 15
Completed | 10 | 13 | 11
Not Completed | 5 | 2 | 4
Not completed — Did not attend the follow up recall | 2 | 2 | 1
Not completed — Failure to comply with the instructions | 3 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Miswak Extract Mouth Wash | Miswak Sticks | Chlorohexidine Gluconate Mouth Wash | Total
Number analyzed (Participants) | 10 | 13 | 11 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 13 | 11 | 34
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 11 | 34
  Male | 0 | 0 | 0 | 0
Self-assessment of mouth odor [Mean (Standard Deviation); unit: units on a scale] — Participants were asked to score their own halitosis on a continuous 10-cm visual analogue scale that is marked as "no odor" on the 0-cm end, and as "extremely foul odor" on the 10-cm end
  units on a scale | 3.70 (3.33) | 3.85 (1.57) | 3.91 (1.3) | 3.83 (2.11)
Organoleptic scores [Mean (Standard Deviation); unit: units on a scale] — Each patient was asked to close her mouth for 3 minutes while breathing only from the nose. Then she was asked to release air from the mouth slowly. The judge kept a distance of about 10 cm between her nose and the patient's mouth to determine the score based on the intensity of the odor.
  The intensity ratings of 0 to 5 score was used where Score 0 stands for "No odor present", score 1 stands "barely noticeable odor", score 2 stands "slight but clearly noticeable odor", score 3 stands "moderate odor", score 4 stands "strong offensive odor" and a Score 5 stands "extremely foul odor"
  units on a scale | 2.6 (0.84) | 2.85 (0.99) | 2.45 (0.69) | 2.65 (0.85)
Volatile sulfur compound [Mean (Standard Deviation); unit: units on a scale] — Scores using breath checker device (Tanita FitScan HC-212SF Breath Checker) were recorded (0=no odor, 1=slight odor, 2=moderate odor, 3=heavy odor, 4=strong odor, 5=intense odor).
  units on a scale | 4.3 (0.48) | 3.15 (1.21) | 4.27 (0.47) | 3.85 (0.99)

OUTCOME MEASURES:

1. Primary Outcome: Organoleptic Scores After the First Use of the Prescribed Method by 15 Minutes (Masking Effect), and After 7 Days of Use (Therapeutic Effect).
Description: The Organoleptic scores were obtained by a calibrated judge who first tested her ability to detect and distinguish odors even at low concentrations using the Smell Identification Test (Sensonics Inc., Haddon Heights, NJ, USA).
  To obtain the score, the patient was asked to close her mouth for approximately 3 minutes while breathing only from the nose. Then he/she was asked to release air from the mouth slowly. The judge kept a distance of about 10 cm between her nose and the patient's mouth to determine the score based on the intensity of the odor.
  The intensity ratings of 0 to 5 score was used where Score 0 stands for "No odor present", score 1 stands "barely noticeable odor", score 2 stands "slight but clearly noticeable odor", score 3 stands "moderate odor", score 4 stands "strong offensive odor" and a Score 5 stands "extremely foul odor".
Time Frame: After the first use of the prescribed method by 15 minutes, and after 7 days of use
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Miswak Extract Mouth Wash | Miswak Sticks | Chlorohexidine Gluconate Mouth Wash
Number analyzed (Participants) | 10 | 13 | 11
units on a scale
  After 15 minutes of first use | 2.10 (1.45) | 1.62 (1.39) | 1.36 (1.03)
  After 7 days of first use | 1.10 (1.20) | 0.54 (0.88) | 1.09 (1.04)
Statistical Analysis 1: Comparison: Miswak Extract Mouth Wash; Paired t-test was performed to examine the significance of change in Organoleptic scores after 15 minutes of the first use of Miswak extract mouth wash; Test type: Superiority or Other; p = 0.299, t-test, 2 sided
Statistical Analysis 2: Comparison: Miswak Extract Mouth Wash; Paired t-test was performed to examine the significance of change in Organoleptic scores after 7 days of using Miswak extract mouth wash; Test type: Superiority or Other; p = 0.007, t-test, 2 sided
Statistical Analysis 3: Comparison: Miswak Sticks; Paired t-test was performed to examine the significance of change in Organoleptic scores after 15 minutes of the first use of Miswak sticks; Test type: Superiority or Other; p = 0.019, t-test, 2 sided
Statistical Analysis 4: Comparison: Miswak Sticks; Paired t-test was performed to examine the significance of change in Organoleptic scores after 7 days of using Miswak sticks; Test type: Superiority or Other; p = 0.000, t-test, 2 sided
Statistical Analysis 5: Comparison: Chlorohexidine Gluconate Mouth Wash; Paired t-test was performed to examine the significance of change in Organoleptic scores after 15 minutes of the first use of Chlorohexidine gluconate mouth wash; Test type: Superiority or Other; p = 0.000, t-test, 2 sided
Statistical Analysis 6: Comparison: Chlorohexidine Gluconate Mouth Wash; Paired t-test was performed to examine the significance of change in Organoleptic scores after 7 days of using Chlorohexidine gluconate mouth wash; Test type: Superiority or Other; p = 0.001, t-test, 2 sided

2. Secondary Outcome: Volatile Sulfur Compound Scores After the First Use of the Prescribed Method by 15 Minutes (Masking Effect), and After 7 Days of Use (Therapeutic Effect)
Description: Scores using breath checker device (Tanita FitScan HC-212SF Breath Checker) were recorded (0=no odor, 1=slight odor, 2=moderate odor, 3=heavy odor, 4=strong odor, 5=intense odor).
Time Frame: After the first use of the prescribed method by 15 minutes, and after 7 days of use
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Miswak Extract Mouth Wash | Miswak Sticks | Chlorohexidine Gluconate Mouth Wash
Number analyzed (Participants) | 10 | 13 | 11
units on a scale
  After 15 minutes of first use | 4.00 (1.25) | 3.38 (0.87) | 4.09 (0.30)
  After 7 days of first use | 3.80 (1.32) | 3.23 (0.73) | 4.00 (0.22)
Statistical Analysis 1: Comparison: Miswak Extract Mouth Wash; Paired t-test was performed to examine the significance of change in Volatile sulfur compound scores after 15 minutes of the first use of Miswak extract mouth wash; Test type: Superiority or Other; p = 0.496, t-test, 2 sided
Statistical Analysis 2: Comparison: Miswak Extract Mouth Wash; Paired t-test was performed to examine the significance of change in Volatile sulfur compound scores after 7 days of using Miswak extract mouth wash; Test type: Superiority or Other; p = 0.244, t-test, 2 sided
Statistical Analysis 3: Comparison: Miswak Sticks; Paired t-test was performed to examine the significance of change in Volatile sulfur compound scores after 15 minutes of the first use of Miswak sticks; Test type: Superiority or Other; p = 0.19, t-test, 2 sided
Statistical Analysis 4: Comparison: Miswak Sticks; Paired t-test was performed to examine the significance of change in Volatile sulfur compound scores after 7 days of of using Miswak sticks; Test type: Superiority or Other; p = 0.829, t-test, 2 sided
Statistical Analysis 5: Comparison: Chlorohexidine Gluconate Mouth Wash; Paired t-test was performed to examine the significance of change in Volatile sulfur compound scores after 15 minutes of the first use of Chlorohexidine gluconate mouth wash; Test type: Superiority or Other; p = 0.341, t-test, 2 sided
Statistical Analysis 6: Comparison: Chlorohexidine Gluconate Mouth Wash; Paired t-test was performed to examine the significance of change in Volatile sulfur compound scores after 7 days of using Chlorohexidine gluconate mouth wash; Test type: Superiority or Other; p = 0.82, t-test, 2 sided

3. Secondary Outcome: Self-assessment of Mouth Odor After 7 Days of Use
Description: Participants were asked to score their own halitosis on a continuous 10-cm visual analogue scale that is marked as "no odor" on the 0-cm end, and as "extremely foul odor" on the 10-cm end
Time Frame: After 7 days of first use
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Miswak Extract Mouth Wash | Miswak Sticks | Chlorohexidine Gluconate Mouth Wash
Number analyzed (Participants) | 10 | 13 | 11
units on a scale | 2.00 (2.16) | 1.92 (1.44) | 2.18 (0.75)
Statistical Analysis 1: Comparison: Miswak Extract Mouth Wash; Paired t-test was performed to examine the significance of change in Self-assessment scores after 7 days of using Miswak extract mouth wash; Test type: Superiority or Other; p = 0.008, t-test, 2 sided
Statistical Analysis 2: Comparison: Miswak Sticks; Paired t-test was performed to examine the significance of change in Self-assessment scores after 7 days of using Miswak sticks; Test type: Superiority or Other; p = 0.001, t-test, 2 sided
Statistical Analysis 3: Comparison: Chlorohexidine Gluconate Mouth Wash; Paired t-test was performed to examine the significance of change in Self-assessment scores after 7 days of using Chlorohexidine gluconate mouth wash; Test type: Superiority or Other; p = 0.02, t-test, 2 sided

ADVERSE EVENTS:
Description: Serious and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Arm/Group | Miswak Extract Mouth Wash | Miswak Sticks | Chlorohexidine Gluconate Mouth Wash
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No